CLINICAL TRIAL: NCT03235349
Title: An Open-Label Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Treatment-Naïve and Treatment-Experienced Asian Adults With Chronic Hepatitis C Virus Genotype (GT) 1 to GT6 Infection With Compensated Cirrhosis and With or Without Human Immunodeficiency Virus Co-Infection
Brief Title: Efficacy and Safety of Glecaprevir/Pibrentasvir (ABT-493/ABT-530) in Treatment-Naive and Treatment-Experienced Asian Adults With Chronic Hepatitis C Virus Genotype (GT) 1 to GT6 Infection With Compensated Cirrhosis and With or Without Human Immunodeficiency Virus Co-Infection
Acronym: VOYAGE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-593
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Chronic Hepatitis C Virus (HCV); Genotype 1 to 6; Cirrhosis; Compensated Cirrhosis; Human Immunodeficiency Virus; co-infection; Treatment-naïve; treatment-experienced; interferon; Asian
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Fibrosis; Acquired Immunodeficiency Syndrome; Coinfection | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glecaprevir/Pibrentasvir (Experimental): Participants received oral glecaprevir/pibrentasvir 300 mg/120 mg once daily (QD) for 12 or 16 weeks. Participants received treatment for 12 weeks with the exception of treatment-experienced, genotype 3-infected participants who received treatment for 16 weeks.
  Interventions: Drug: Glecaprevir/Pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir — Coformulated tablet for oral administration
  Other Names: ABT-493/ABT-530; MAVYRET™

SUMMARY:
This study will evaluate the efficacy and safety of glecaprevir/pibrentasvir (ABT-493/ABT-530) in chronic hepatitis C virus (HCV) genotype (GT)1 to GT6-infected Asian participants with compensated cirrhosis with or without human immunodeficiency virus (HIV) co-infection who are HCV treatment-naïve or treatment-experienced with interferon (IFN) (alpha, beta or pegylated interferon [pegIFN]) with or without ribavirin (RBV) OR sofosbuvir with RBV with or without IFN.

ELIGIBILITY:
Inclusion Criteria:

* Must be of Asian descent.
* Screening laboratory result indicating hepatitis C virus (HCV) genotype (GT) 1, 2, 3, 4, 5 or 6 infection.
* Positive anti-HCV antibody (Ab) and HCV ribonucleic acid (RNA) greater than or equal to 1000 IU/ mL at Screening Visit.
* Chronic HCV infection defined as one of the following:

  * Positive for anti-HCV Ab or HCV RNA at least 6 months before Screening; or
  * A liver biopsy consistent with chronic HCV infection;
* HCV treatment-naïve to any approved or investigational HCV treatment or treatment-experienced with interferon (IFN) (alpha, beta or pegylated interferon [pegIFN] with or without ribavirin (RBV) OR sofosbuvir with RBV with or without IFN. Previous treatment must have been completed >= 8 weeks prior to screening.
* Compensated cirrhosis defined as Child-Pugh score of ≤ 6 at Screening and no current or past clinical evidence of Child-Pugh B or C Classification or clinical history of liver decompensation including ascites noted on physical exam, bleeding varices, use of diuretics for ascites, or hepatic encephalopathy.
* Absence of hepatocellular carcinoma (HCC)

Participants enrolled with human immunodeficiency virus (HIV)-1 and HCV co-infection must also meet the following criteria:

* Positive test result for human immunodeficiency virus antibody (HIV Ab) at Screening.
* Naïve to treatment with any antiretroviral therapy (ART) with a cluster of differentiation (CD)4+ count greater than or equal to 500 cells/mm³ (or CD4+ % >= 29%), or
* On a stable, qualifying HIV-1 ART regimen with CD4+ count >= 200 cells/mm³ (or CD4+ % >= 14%) at Screening; and plasma HIV-1 RNA below lower limit of quantification (LLOQ) by an approved plasma HIV-1 RNA quantitative assay at Screening and at least once during the 12 months prior to Screening.

Exclusion Criteria:

* Positive test result for hepatitis B surface antigen (HbsAg) or positive test result for hepatitis B virus (HBV) deoxyribonucleic acid (DNA) if HBsAg is negative.
* Any cause of liver disease other than chronic HCV-infection.
* HCV genotype performed during screening indicating co-infection with more than one HCV genotype
* Clinically significant abnormalities, other than HCV infection or HCV/HIV co-infection
* Chronic human immunodeficiency virus, type 2 (HIV-2) infection

Additional Exclusion Criteria for participants with HCV/HIV Co-Infection:

* For participants on stable ART, taking anti-retroviral agent(s) other than those permitted
* Treatment for an acquired immunodeficiency syndrome (AIDS)-associated opportunistic infection within 12 months of Screening or prophylaxis for an AIDS-associated opportunistic infection within 6 months of screening
* Diagnosis of any clinical AIDS-defining event within 12 months prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (34):
- China (25):
  - Peking University Peoples Hospit /ID# 156851, Beijing, Beijing Municipality
  - Guangzhou Eighth People's Hosp /ID# 156865, Guangzhou, Guangdong
  - Guangdong General Hospital /ID# 156827, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 156866, Guangzhou, Guangdong
  - The Third Affiliated Hospital Of Sun Yat-Sen University /ID# 156905, Guangzhou, Guangdong
  - The Second Hospital of Nanjing /ID# 156869, Nanjing, Jiangsu
  - Jiangsu Province People's Hospital /ID# 156867, Nanjing, Jiangsu
  - The First Hosp of Jilin Univ /ID# 156825, Changchun, Jilin
  - The Sixth People's Hospital of Shenyang /ID# 156854, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong /ID# 157337, Shanghai, Shanghai Municipality
  - Huashan Hospital of Fudan University /ID# 156909, Shanghai, Shanghai Municipality
  - Shanghai Public Health Cli Ctr /ID# 156837, Shanghai, Shanghai Municipality
  - West China Hospital /ID# 156835, Chengdu, Sichuan
  - Beijing Di Tan Hospital, Capital Medical University /ID# 156852, Beijing
  - 1st Hospital of Peking Uni /ID# 156850, Beijing
  - Beijing Friendship Hospital /ID# 156843, Beijing
  - Beijing Youan Hosp, Cap Med Un /ID# 163418, Beijing
  - 2nd Affiliated Hosp Chongqing /ID# 156838, Chongqing
  - Mengchao Hepatobiliary Hospita /ID# 156907, Fuzhou
  - Chinese People's Liberation Army 81 Hospital /ID# 156868, Nanjing
  - Shengjing Hospital of China Medical University /ID# 156829, Shenyang
  - 1st Aff Hosp Xinjiang Med Uni /ID# 156891, Ürümqi
  - Fourth Military Medical University Tangdu Hospital, PLA /ID# 156767, Xi'an
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University /ID# 163420, Xi'an
  - Henan Provincial Peoples Hosp /ID# 157371, Zhengzhou, Henan
- South Korea (9):
  - Pusan National University Hosp /ID# 163411, Busan, Busan Gwang Yeogsi
  - Seoul National Univ Bundang ho /ID# 163408, Seongnam, Gyeonggido
  - Inje University Busan Paik Hospital /ID# 163384, Pusan, Gyeongsangbuk-do
  - Pusan Nat Univ Yangsan Hosp /ID# 163385, Yangsan, Gyeongsangnam-do
  - Severance Hospital /ID# 163399, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 163402, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 163412, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 163401, Seoul
  - Asan Medical Center /ID# 163398, Seoul

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Wei L, Wang G, Alami NN, Xie W, Heo J, Xie Q, Zhang M, Kim YJ, Lim SG, Fredrick LM, Lu W, Liu W, Kalluri HV, Krishnan P, Tripathi R, Mobashery N, Burroughs M, Asatryan A, Jia J, Hou J. Glecaprevir-pibrentasvir to treat chronic hepatitis C virus infection in Asia: two multicentre, phase 3 studies- a randomised, double-blind study (VOYAGE-1) and an open-label, single-arm study (VOYAGE-2). Lancet Gastroenterol Hepatol. 2020 Sep;5(9):839-849. doi: 10.1016/S2468-1253(20)30086-8. Epub 2020 Jul 16. PMID 32682494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 34 sites in China and South Korea. Eligible participants were chronic hepatitis C (HCV) genotype (GT)1-6-infected adults with compensated cirrhosis with or without HIV co-infection who were HCV treatment-naïve or treatment-experienced with regimens containing interferon (IFN), pegylated IFN, ribavirin, and/or sofosbuvir.
Period: Overall Study
Arm/Group | Glecaprevir/Pibrentasvir
Started | 160
Completed | 158
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.83 (11.27)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 120
  ≥ 65 years | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 160
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 37
  China | 123
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 85
  Genotype 2 | 53
  Genotype 3 | 14
  Genotype 4 | 1
  Genotype 5 | 0
  Genotype 6 | 7
Prior HCV Treatment History [Count of Participants; unit: Participants] — Treatment-experienced includes treatment with interferon (IFN; alpha, beta or pegylated interferon [pegIFN]) with or without ribavirin (RBV), OR sofosbuvir with RBV with or without IFN.
  Participants
    Treatment-naive | 110
    Treatment-experienced | 50
HCV Ribonucleic Acid (RNA) Level [Mean (Standard Deviation); unit: log₁₀ IU/mL] | 6.16 (0.74)
Human Immunodeficiency Virus (HIV) Co-infection Status [Count of Participants; unit: Participants]
  Hepatitis C infection only | 160
  HCV / HIV co-infection | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (LLOQ; 15 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug, Week 24 or Week 28 depending on the treatment regimen.
Population: All enrolled participants who received at least 1 dose of study drug. Backward imputation, where applicable, was used to impute missing data. Participants with missing data after backward imputation were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 160
percentage of participants | 99.4 [98.2 to 100.0]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as meeting one of the following:
  * confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements > 1 log₁₀ IU/mL above nadir) at any time point during the treatment period; or
  * confirmed HCV RNA greater than or equal to 100 IU/mL after HCV RNA < 15 IU/mL during the treatment period, or
  * HCV RNA ≥ 15 IU/mL at end of treatment with at least 6 weeks of treatment.
Time Frame: 12 or 16 weeks depending on the treatment regimen
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 160
percentage of participants | 0.0 [0.0 to 2.3]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA greater than or equal to 15 IU/mL between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < 15 IU/mL at the end of treatment, excluding re-infection.
Time Frame: From the end of treatment (Week 12 or 16) through 12 weeks after the last dose of study drug (Weeks 24 or 28 depending on the treatment regimen).
Population: All enrolled participants who received at least one dose of study drug, with HCV RNA < 15 IU/mL at the end of treatment, at least one post-treatment HCV RNA value, and who completed the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 159
percentage of participants | 0.6 [0.1 to 3.5]

4. Secondary Outcome: Percentage of HCV/HIV Co-infected Participants Achieving SVR12
Description: SVR12 was defined as plasma HCV RNA level less than LLOQ (15 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug, Week 24 or Week 28 depending on the treatment regimen
Population: No HCV-HIV co-infected participants were enrolled in the study
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From initiation of study drug through 30 days after last dose; up to 16 or 20 weeks depending on the treatment regimen.
Arm/Group | Glecaprevir/Pibrentasvir
All-Cause Mortality (participants affected / at risk) | 1/160
Serious Adverse Events (participants affected / at risk) | 5/160
Other Adverse Events (participants affected / at risk) | 29/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=160)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1)
HEPATIC LESION (Hepatobiliary disorders) | 1 (1)
LIVER ABSCESS (Infections and infestations) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=160)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 19 (19)
URINARY TRACT INFECTION (Infections and infestations) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT03235349/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT03235349/SAP_001.pdf